CLINICAL TRIAL: NCT03727997
Title: Epidemiology and Long Term Outcome of Critically Ill Patients Requiring Renal Replacement Therapy in Southeast Asia and India (InSEA-RRT Registry)
Acronym: InSEA-RRT
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Faculty of Medicine, Chulalongkorn University
Other Study IDs: InSEA-RRT Registry
Record Dates: First submitted 2018-10-26; First posted 2018-11-01 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Renal replacement therapy; Intensive Care Unit
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AKI patients stage 3

SUMMARY:
Acute kidney injury is associated with increased short-term and long-term morbidity and mortality. Long-term data is lacking in low to middle-income countries. Our study aims to follow the acute kidney injury patients stage 3 in intensive care units for 2 years to observe mortality and associated factors.

ELIGIBILITY:
Inclusion Criteria:

* AKI stage 3
* At least 18 years old

Exclusion Criteria:

* ESRD patients (eGFR < 15 mL/min/1.73 m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted in intensive care units who are diagnosed with acute kidney injury by KDIGO criteria (cr or urine output criteria) stage 3
Sampling Method: Non-Probability Sample
Enrollment: 2315 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
2-year mortality | 2-year

SECONDARY OUTCOMES:
Hospital mortality | 28-day
RRT rate | 28-day
Renal recovery | 28-day
  Number of Participants with who survive. Number of Participants with dialysis independence and creatinine <1.5 mg/dL
2-year major adverse kidney events | 2-year
  Number of Participants with 25% or greater decline in eGFR. Number of participants who receive new renal replacement therapy (RRT).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Pathumwan, Thailand

IPD SHARING:
Plan to Share IPD: No